CLINICAL TRIAL: NCT04030832
Title: Reconstruction of Skin Substance Loss With Method of "Micro-grafts" Obtained by Mechanical Disintegration: Preliminary Study
Brief Title: Reconstruction of Skin Substance Loss With "Micro-grafts" Obtained by Mechanical Disintegration
Acronym: MG-1
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Michele Riccio, Director, Azienda Ospedaliero, Universitaria Ospedali Riuniti
Other Study IDs: MICROINNESTI-1
Record Dates: First submitted 2019-07-17; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Cutaneous Ulcer; Trauma Injury
MeSH Terms: conditions — Skin Ulcer; Accidental Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The etiology of non-healing ulcers depends on both systemic and local factors. The introduction of advanced dressing, negative wound therapy and compression therapy have undoubtedly improved clinical outcomes. The principal aim of study was to demonstrate the efficacy of skin micrografts in the treatment of skin substance loss.

DETAILED DESCRIPTION:
The principal aim of study was to evaluate the efficacy of skin micro-grafts obtained with the system of mechanical disintegration in the reconstruction of skin substance loss in the limbs.

The primary endpoint consists in evaluating, through a specific evaluation scale, the Wound Bed Score (WBS) for skin substance loss at Time 0 (T0) and 30 days after the procedure (T30) and to evaluate the increase of this score in this time frame set at 50%. The evaluation will be carried out in double blind.

The secondary endpoints instead consist in the evaluation of the Wound Surface Area Assessment to be carried out at T0 and T30.

In the evaluation of the quality of the resulting scars, through the Vancouver Scale (VS), 90 (T90) and 180 days (T180) after treatment and to evaluate the reduction of this score by 15%; on the other in the evaluation of the progress of the Visual Analogic Scale (VAS) administered to the patient at T0, 30, 90, 180.

The purpose of this minimally invasive treatment is to improve the quality of life of those affected by these injuries, avoiding the use of prolonged advanced medications and / or more invasive surgical procedures, thus speeding up healing and favoring the clinical outcome of patients.

No chemical reagents or enzymes are used for the method. There is therefore no tissue manipulation, in full compliance with the European directive 23/2004.

ELIGIBILITY:
Inclusion Criteria:

* Full-thickness skin loss from a minimum size of 3x3 cm (9cm2) to a maximum size of 5x5 cm (25cm2);
* Loss of substance caused by abrasive-contusive traumas (loss of full-thickness skin substance) or by thermal burn (deep degree II), present for at least 15 days;
* Absence of clinical signs of infection assessed by two culture swabs performed at T0 (pre and post debridement);
* Pre-operative inflammatory index (VES, PCR) and b-hcg negative;
* Absence of exposure of osteo-cartilaginous structures, of noble structures (major arterial vessels, major nerve trunks, tendons without paratenon);
* Specific written informed consent

Exclusion Criteria:

* Smoking patients (≥ 10 cigarettes / day);
* Patients with type I or type II diabetes mellitus:
* Patients suffering vascular trophic ulcers;
* Patients with loss of substance at the level of the fingers and toes;
* Patients with loss of substance of the foot and the yarrow region;
* Patients with oncological pathologies in progress or in remission;
* Patients in therapy with immunosuppressive and corticosteroid drugs, anticoagulants, antiplatelet agents;
* Patients with autoimmune diseases including connectivitis;
* Patients with congenital, acquired and metabolic immunodeficiencies;
* Pregnant patients (ascertained with β-HCG) and breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attend the various regional hospitals through the emergency room or surgical clinic
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Wound Bed Score values | change of baseline wound bed score values at day 30
  Percentage of patients with change of the Wound Bed Score values higher than 50%, after 30 days,

SECONDARY OUTCOMES:
Spontaneous re-epithelialization. | Day 0 and Day 30
  Percentage of patients with spontaneous re-epithelialization of the total wound surface, after 30 days, as assessed by Wound Surface Area Assessment
Vancouver scale | Day 30, Day 90 and Day 180
  Percentage of patients with change of Vancouver scale values higher than 15%

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria Ospedali Riuniti, Ancona, AN
  - IRCCS Policlinico San Donato, Milan, MI
  - Università degli Studi di Udine, Udine, UD
  - Università degli Studi di Roma "La Sapienza", Roma

REFERENCES:
- [Result] Greaves NS, Ashcroft KJ, Baguneid M, Bayat A. Current understanding of molecular and cellular mechanisms in fibroplasia and angiogenesis during acute wound healing. J Dermatol Sci. 2013 Dec;72(3):206-17. doi: 10.1016/j.jdermsci.2013.07.008. Epub 2013 Jul 30. PMID 23958517
- [Result] Trovato L, Monti M, Del Fante C, Cervio M, Lampinen M, Ambrosio L, Redi CA, Perotti C, Kankuri E, Ambrosio G, Rodriguez Y Baena R, Pirozzi G, Graziano A. A New Medical Device Rigeneracons Allows to Obtain Viable Micro-Grafts From Mechanical Disaggregation of Human Tissues. J Cell Physiol. 2015 Oct;230(10):2299-303. doi: 10.1002/jcp.24973. PMID 25728337
- [Result] Marcarelli M, Trovato L, Novarese E, Riccio M, Graziano A. Rigenera protocol in the treatment of surgical wound dehiscence. Int Wound J. 2017 Feb;14(1):277-281. doi: 10.1111/iwj.12601. Epub 2016 Apr 29. PMID 27126653
- [Result] Baglioni E, Trovato L, Marcarelli M, Frenello A, Bocchiotti MA. Treatment of Oncological Post-surgical Wound Dehiscence with Autologous Skin Micrografts. Anticancer Res. 2016 Mar;36(3):975-9. PMID 26976986
- [Result] Svolacchia F, De Francesco F, Trovato L, Graziano A, Ferraro GA. An innovative regenerative treatment of scars with dermal micrografts. J Cosmet Dermatol. 2016 Sep;15(3):245-53. doi: 10.1111/jocd.12212. Epub 2016 Jan 30. PMID 26825041
- [Result] De Francesco F, Graziano A, Trovato L, Ceccarelli G, Romano M, Marcarelli M, Cusella De Angelis GM, Cillo U, Riccio M, Ferraro GA. A Regenerative Approach with Dermal Micrografts in the Treatment of Chronic Ulcers. Stem Cell Rev Rep. 2017 Feb;13(1):139-148. doi: 10.1007/s12015-016-9692-2. PMID 27738884
- [Result] Falanga V, Saap LJ, Ozonoff A. Wound bed score and its correlation with healing of chronic wounds. Dermatol Ther. 2006 Nov-Dec;19(6):383-90. doi: 10.1111/j.1529-8019.2006.00096.x. PMID 17199681
- [Result] Qi X, Ding L, Huang W, Wen B, Guo X, Zhang J. An improved automated type-based method for area assessment of wound surface. Wound Repair Regen. 2017 Jan;25(1):150-158. doi: 10.1111/wrr.12495. Epub 2017 Jan 25. PMID 27859908
- [Result] Baryza MJ, Baryza GA. The Vancouver Scar Scale: an administration tool and its interrater reliability. J Burn Care Rehabil. 1995 Sep-Oct;16(5):535-8. doi: 10.1097/00004630-199509000-00013. PMID 8537427
- [Result] Jimi S, Kimura M, De Francesco F, Riccio M, Hara S, Ohjimi H. Acceleration Mechanisms of Skin Wound Healing by Autologous Micrograft in Mice. Int J Mol Sci. 2017 Aug 2;18(8):1675. doi: 10.3390/ijms18081675. PMID 28767054